CLINICAL TRIAL: NCT06770231
Title: Peri-implant Bone Behavior After Single Drilling Technique Versus Undersized Technique of Immediately Loaded Implant in Posterior Maxilla: A One-year Prospective Study
Brief Title: Peri-implant Bone Behaviour Using Two Drilling Techniques in Posterior Maxilla
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Galal, Clinical demonstrator oral and maxillofacial surgery Mansoura university, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A03012024OS
Record Dates: First submitted 2025-01-01; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Implant
Keywords: Implant stability; Immediate loading; Single drilling technique; Posterior maxilla

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Undersized technique (Experimental): New drilling tech
  Interventions: Other: Single drill system
- Single drill technique (Active Comparator): One drill system
  Interventions: Other: Single drill system

INTERVENTIONS:
Other: Single drill system — New system for drilling

SUMMARY:
Two different drilling techniques in posterior maxilla immediate loading implant

DETAILED DESCRIPTION:
One of the surgical techniques used to enhance the primary stability of implant in low density bone was the undersized drilling technique, which has been introduced to locally optimize poor density of bone by using a final drill diameter considerably smaller compared with the implant diameter.

On the other hand, a novel hollow drill with a single drilling systems was designed. Single drilling technique shortens surgical times, removes the smallest amount of bone during implant site preparation, reduces bone damage and micro fractures, and speeds up the healing process. Additionally, because of the hollow shape, bone core may be harvested and used as an autogenous bone grafting material.

ELIGIBILITY:
Inclusion criteria:

1. Patients with missing single or multiple teeth in posterior maxilla.
2. Age more than 18 years.
3. 10 mm or more vertical bone height is present.
4. Good oral hygiene.
5. Patients willing to be present during the study follow up intervals.
6. Patients free from any systemic diseases.
7. 6 mm or more ridge width is present.
8. Crown height space of at least 8 mm.
9. Patients without any para-functional habits (bruxism and clenching).

Exclusion criteria:

1. Patients with any pathological lesion or root tips at the planned surgical site.
2. Patients with inadequate bone height and thickness.
3. Smoking more than 14 cigarettes per day.14
4. Alcohol or drug abuse.
5. Patients with systemic diseases that absolutely contraindicate implant placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Implant stability | 12 months
  Implant stability will be assessed at the time of implant insertion and at 3, 6 and 12 months after surgery.
Modified Sulcus Bleeding Index (mBI) | 12 months
  It will be measured at 3,6 and 12 months post-operatively. Clinical signs and symptoms of inflammation of peri-implant mucosa will be graded using criteria of modified sulcus bleeding index (mBI).
Peri-implant probing depth | 12 months
  Depth of the peri-implant sulcus will be recorded initially at the time of loading, 3, 6 and 12 months following implant loading by a graduated periodontal probe with light force to avoid undue tissue damage and over-extension into the healthy tissue
Marginal Bone Loss | 12 months
  For the calculation of marginal bone loss (MBL), the implant will be used as a reference by adjusting the cross-sectional and panoramic long axis in the center of the implant and bisecting it
Bone Density Recordings | 12 months
  Relative bone density records will be collected from the bucco-palatal view of the cross-sectional plane using the greyscale bone measuring tool

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Two groups one single drill and undersized groups with 12 months follow up
Supporting Information: Study Protocol
Time Frame: 12 month
Access Criteria: All

REFERENCES:
- [Derived] Sadek MAG, Amer MZ, El-Gohary N, Elsheikh HA. Peri-implant bone behavior after single drilling technique versus undersized drilling technique of immediately loaded implant in posterior maxilla: a one-year prospective study. BMC Oral Health. 2025 Jun 21;25(1):956. doi: 10.1186/s12903-025-06360-0. PMID 40544298